CLINICAL TRIAL: NCT03894787
Title: Ross for Valve Replacement in AduLts (REVIVAL) Registry
Brief Title: Ross for Valve Replacement in Adults - Registry
Acronym: REVIVAL-Reg
Status: Completed | Type: Observational
Sponsor: Population Health Research Institute (Other)
Collaborators: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Other Study IDs: REVIVAL Reg - 2018
Record Dates: First submitted 2019-03-22; First posted 2019-03-29 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Aortic Valve Disease
Keywords: Ross procedure; Conventional aortic valve replacement
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This registry follows patients undergoing two methods of aortic heart valve replacement in adults aged 18-60, the Ross procedure or conventional aortic valve replacement using a biologic or mechanical heart valve. The Ross procedure replaces a patient's diseased aortic valve with his/her own pulmonary valve and uses a donor valve in the pulmonary position which receives less stress than the aortic valve. Mechanical valves tend to form blood clots so they need long-term blood thinners that increase risk of bleeding and lower quality of life. Animal tissue valves reduce clotting and bleeding risks but wear out sooner and shorten patient life-span. The REVIVAL Registry will run in parallel with the REVIVAL randomized trial.

DETAILED DESCRIPTION:
Heart valves help control blood flow through the heart and, if diseased, may need to be replaced. After having a heart valve replaced, patients have a higher risk of death than people who have not had a valve replaced. In young adult patients, replacing the aortic heart valve with a mechanical valve halves their life-span compared to other people their age. Mechanical valves tend to form blood clots so they need long-term blood thinners that increase risk of bleeding and lower quality of life. Animal tissue valves reduce clotting and bleeding risks but wear out sooner and shorten patient life-span. An operation, called the Ross procedure, replaces a patient's diseased aortic valve with his/her own pulmonary valve and uses a donor valve in the pulmonary position which receives less stress than the aortic valve. The Ross procedure aims to improve valve durability with less clotting, avoiding use of blood thinners. Patients and physicians need a large, high-quality study comparing the Ross procedure and standard valve replacement to know if either approach is better. In parallel to the REVIVAL Registry, a REVIVAL Randomized Trial will also take place.

Patients included in randomized trials often systematically differ from those who are not. By creating a registry of patients who are eligible for but not recruited into the REVIVAL trial, the investigators will better understand: 1) the reasons for not including these patients; 2) how those patients differ in terms of baseline characteristics from the trial cohort; 3) whether the outcomes of registry participants differ from those in the trial, assessed by treatment group. The registry will aid in understanding the generalizability of the results that the trial produces.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60 years
2. Undergoing clinically indicated aortic valve replacement
3. Provided written informed consent

Exclusion Criteria:

1. Previous valve replacement not in the aortic position
2. Patients undergoing concomitant CABG or other valve procedure during aortic valve replacement
3. Known connective tissue disease
4. Severe (grade 3 or 4) right or left ventricular dysfunction
5. Pulmonary valve dysfunction or anomaly not compatible with the Ross procedure (as determined by the consulting cardiac surgeon)
6. Life expectancy less than 5 years (as determined by the consulting cardiac surgeon)
7. Documented severe aortic insufficiency not solely due to leaflet issue
8. Previous intervention on the pulmonary valve

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All patients who meet eligibility criteria of the REVIVAL trial, but are not included in the trial due to patient or clinician factors, will be asked to participate in the REVIVAL registry.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Evaluation of systematic differences between registry and trial patients | Through REVIVAL Trial completion, estimated to be 10 years
  The primary outcome of the REVIVAL registry is to examine for systematic differences between the demographics and outcomes of patients enrolled in the REVIVAL trial and patients not enrolled in the trial.
  We will use descriptive statistics including mean (standard deviation), median (interquartile range), and count (proportion) to describe the REVIVAL registry cohort.

SECONDARY OUTCOMES:
Evaluate the number of patients meeting eligibility criteria for the REVIVAL trial per month who are not enrolled into the trial. | Through completion of the pilot trial, estimated to be 3 years
  To determine the number of eligible patients and reasons why they were not enrolled into the REVIVAL trial.
Evaluate the proportion of Ross procedures compared to conventional aortic valve replacement. | Through completion of the pilot trial, estimated to be 3 years
  Measure the proportions of type of mechanical valve versus biological valves versus Ross procedure in the REVIVAL registry participants.
The rate of survival free of a composite of life-threatening valve-related complications (major bleeding, stroke or systemic thromboembolism, valve thrombosis, and operated-on valve reintervention) | Through trial completion, estimated to be 10 years
  Evaluate the frequency of REVIVAL trial outcomes among registry participants.
  The primary outcome is the rate of survival free of life-threatening valve-related complications (major bleeding, stroke or systemic thromboembolism, valve thrombosis, and operated-on valve reintervention) over duration of follow-up. Assessment of this composite over time is particularly important, as the Ross procedure may show initial benefit secondary to thromboembolic and bleeding reduction, however should the technique show high late rates of reoperation as suggested in some observational literature, the effect magnitude may change significantly over time.
The rate of perioperative and non-perioperative major bleeding over the duration of patient follow-up. | Through trial completion, estimated to be 10 years
  Evaluate the frequency of REVIVAL trial outcomes among REVIVAL registry participants.
  Perioperative (index surgery only) Intraoperative: After administration of protamine, delay of chest closure for bleeding > 500 mL/hr requiring packing and transfusion of more than 3 units red blood cells /whole blood.
  Upon leaving OR to 48hrs postop (modified BARC type 4)
  Intracranial bleeding within 48hrs Reoperation after sternum closure for purpose of controlling bleeding or relief of tamponade Transfusion of ≥ 5 units packed red blood cells /whole blood in the 48hr period Chest tube output ≥ 2L in the first 24hr Non-perioperative Per the International Society of Thrombosis and Hemostasis (ISTH) major bleeding definition.
The rate of stroke or systemic thromboembolism over the duration of patient follow-up. | Through trial completion, estimated to be 10 years
  Evaluate the frequency of REVIVAL trial outcomes among REVIVAL registry participants.
  Stroke is acute focal brain dysfunction due to a vascular cause lasting ≥ 24 hrs in the absence of brain imaging or requires evidence of acute stroke on brain imaging. Stroke is divided into 3 types: ischemic stroke, hemorrhagic stroke, and undetermined stroke. If death occurs within 24 hours, the neurological deficit must persist up to the time of death.
  Systemic arterial embolism is an abrupt vascular insufficiency associated with evidence of arterial occlusion in the absence of other likely mechanisms. Clinical signs/symptoms must be consistent with embolic arterial occlusion, there must be clear evidence of abrupt occlusion of a systemic artery, with at least one type of supporting evidence (surgical report indicating evidence of arterial embolism, pathological specimens related to embolism removal, imaging evidence consistent with arterial embolism, or autopsy report).
The rate of valve thrombosis per VARC criteria over the duration of patient follow-up. | Through trial completion, estimated to be 10 years
  Evaluate the frequency of REVIVAL trial outcomes among REVIVAL registry participants.
  Valve thrombosis is defined as any thrombus not caused by infection attached to or near an operated valve that occludes part of the blood flow path, interferes with valve function, or is large enough to warrant treatment. Valve thrombus found at autopsy in a patient whose cause of death was not valve related or found at operation for and unrelated indication is to be counted as valve thrombosis.
The rate of operated-on valve reintervention over the duration of patient follow-up. | Through trial completion, estimated to be 10 years
  Evaluate the frequency of REVIVAL trial outcomes among REVIVAL registry participants.
  Rate of valve reintervention Any surgical or percutaneous procedure that repairs, or otherwise alters or adjusts, or replaces a previously implanted prosthesis or valve.
Rate of mortality within 30 days post-operatively. | 30 days
  Evaluate the frequency of REVIVAL trial outcomes among REVIVAL registry participants.
Measure health related quality of life using the 36-Item Short Form Survey (SF-36) questionnaire over the duration of patient follow-up | Through trial completion, estimated to be 10 years
  Evaluate the frequency of REVIVAL trial outcomes among REVIVAL registry participants.
  The 36-Item Short Form Survey (SF-36) is a health related quality of life questionnaire that measure eight health domains and each survey provides psychometrically-based physical component summary (PCS) and mental component summary (MCS) scores. The domains are physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. The questionnaire is calibrated such that scored values of 50 represent the norm and higher scored values according to the scoring key represent a more favourable health state. A baseline score will be obtained prior to the patient's surgery and the SF-36 will be administered annually thereafter over the duration of patient follow-up.
The rate of operated-valve endocarditis over the duration of patient follow-up | Through trial completion, estimated to be 10 years
  Evaluate the frequency of REVIVAL trial outcomes among REVIVAL registry participants.
  Defined as any infection involving a valve on which an operation has been performed. The diagnosis is based on one or more of the following: 1) reoperation with evidence of abscess, paravalvular leak, pus, or vegetation confirmed as secondary to infection by histologic or bacteriologic studies; 2) autopsy findings of abscess, pus, or vegetation involving an operated-on valve; or 3) the meeting of Duke criteria for endocarditis.
The rate of aortic valve re-intervention over the duration of patient follow-up. | Through trial completion, estimated to be 10 years
  Evaluate the frequency of REVIVAL trial outcomes among REVIVAL registry participants
  Any surgical or percutaneous procedure that repairs, or otherwise alters or adjusts, or replaces a previously implanted prosthesis or valve in the aortic position.
The rate of pulmonary valve re-intervention over the duration of patient follow-up. | Through trial completion, estimated to be 10 years
  Evaluate the frequency of REVIVAL trial outcomes among REVIVAL registry participants
  Any surgical or percutaneous procedure that repairs, or otherwise alters or adjusts, or replaces a previously implanted prosthesis or valve in the pulmonary position.
Mean aortic valve gradient. | Through trial completion, estimated to be 10 years
  Evaluate the frequency of REVIVAL trial outcomes among REVIVAL registry participants.
  Measured through echocardiography
Mean pulmonic valve gradient | Through trial completion, estimated to be 10 years
  Evaluate the frequency of REVIVAL trial outcomes among REVIVAL registry participants.
  Measured through echocardiography
Severity of aortic valve regurgitation. | Through trial completion, estimated to be 10 years
  Evaluate the frequency of REVIVAL trial outcomes among REVIVAL registry participants.
  Measured through echocardiography, categorized as mild, moderate, or severe
Severity of pulmonic valve regurgitation | Through trial completion, estimated to be 10 years
  Evaluate the frequency of REVIVAL trial outcomes among REVIVAL registry participants.
  Measured through echocardiography, categorized as mild, moderate, or severe

OTHER OUTCOMES:
Rate of myocardial infarction | 30 days postoperatively
  Myocardial infarction (Fourth universal definition)
  Occurring after 48 hrs post-operative, clinical evidence of acute myocardial injury with detection of a rise and/or fall of cTn values with at least one value above the 99th percentile URL and at least one of:
  Symptoms of myocardial ischemia New ischemic ECG changes Development of pathological Q waves Imaging evidence of new loss of viable myocardium or a new regional wall motion abnormality in a pattern consistent with an ischemic etiology; indication of a coronary thrombus by angiography or autopsy.
Rate of acute renal failure by Acute Kidney Injury Network classification | 30 days postoperatively
  Acute renal failure By AKIN classification - An abrupt (within 48 hours) reduction in kidney function currently defined as an absolute increase in serum creatinine of more than or equal to 0.3 mg/dl (≥ 26.4 μmol/l), a percentage increase in serum creatinine of more than or equal to 50% (1.5-fold from baseline), or a reduction in urine output (documented oliguria of less than 0.5 ml/kg per hour for more than six hours).
Rate of need for acute renal replacement therapy | 30 days postoperatively
  The rate of patients requiring new renal replacement therapy within 30 days of surgery.
Rate of surgical re-exploration of the mediastinum for bleeding | 30 days postoperatively
  Surgical re-exploration of the mediastinum for bleeding
Rate of deep mediastinal wound infection | 30 days postoperatively
  Deep mediastinal wound infection

CONTACTS AND LOCATIONS:
Overall Officials: Richard Whitlock, MD, PhD, Principal Investigator — Population Health Research Institute
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada